CLINICAL TRIAL: NCT06677684
Title: The Effect of Adjunct Vitamin a on Community-Acquired Pneumonia in Southern Iranian Children: a Randomized Clinical Trial
Acronym: CAP Vitamin A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Bagher Rahmati, Facualty memeber Oh HUMS, Hormozgan University of Medical Sciences
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: IR.HUMS.REC.1400.113
Record Dates: First submitted 2024-11-01; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2021-02

CONDITIONS: Community-Acquired Pneumonia; Vitamin a
Keywords: Community-acquired pneumonia; Vitamin A; Pediatrics; Hospitalization; Southern Iran
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Vitamin A

STUDY DESIGN:
Intervention Model Description: This randomized clinical trial included 105 children with CAP who were admitted to Bandar Abbas Children's Hospital. Participants were randomly assigned to two groups: a control group receiving standard antibiotic therapy and an intervention group receiving standard antibiotics plus vitamin A (25,000 IU for 2 days).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- a control group (No Intervention): the control group received standard antibiotic therapy
- the intervention group received standard antibiotics plus adjunctive vitamin A supplementation (Experimental): the intervention group received standard antibiotics plus adjunctive vitamin A supplementation (25,000 IU daily for two days)
  Interventions: Dietary Supplement: Vitamin A

INTERVENTIONS:
Dietary Supplement: Vitamin A — the intervention group received standard antibiotics plus adjunctive vitamin A supplementation (25,000 IU daily for two days)
  Arms: the intervention group received standard antibiotics plus adjunctive vitamin A supplementation

SUMMARY:
This randomized clinical trial included 105 children with CAP who were admitted to Bandar Abbas Children's Hospital. Participants were randomly assigned to two groups: a control group receiving standard antibiotic therapy and an intervention group receiving standard antibiotics plus vitamin A (25,000 IU for 2 days). Key data collected included age, sex, duration of hospitalization, treatment duration, and daily Respiratory Index of Severity in Children (RISC) scores.

DETAILED DESCRIPTION:
Children to present with CAP symptoms

ELIGIBILITY:
Inclusion Criteria:

* children to present with CAP symptoms, including fever, cough, pulmonary rales, respiratory distress (age-adjusted tachypnea: >50 breaths per minute for infants under 1 year, >40 for ages 1-5 years, and >30 for those over 5 years), and radiographic findings indicative of pneumonia.

Exclusion Criteria:

* underlying immunodeficiency, chronic respiratory conditions, concurrent use of immunosuppressive medications, prior high-dose vitamin A intake, and hospitalizations shorter than 24 hours

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 105 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-18 (Actual)

PRIMARY OUTCOMES:
duration of hospitalization | Key data collected included age, sex, duration of hospitalization, treatment duration, and daily Respiratory Index of Severity in Children (RISC) scores.
  Vitamin A supplementation was associated with a significant reduction in hospitalization duration in children with CAP, supporting its potential as an adjunct therapy.
Treatment duration daily Respiratory Index of Severity in Children (RISC) scores | From enrollment to the end of treatment and discharge of patients ( 6 months)
  daily Respiratory Index of Severity in Children (RISC) scores

CONTACTS AND LOCATIONS:
Locations (1):
- Hormozgan University of Medical Sciences, Bandar Abbas, Hormozgan, Iran

IPD SHARING:
Plan to Share IPD: Undecided